CLINICAL TRIAL: NCT01805271
Title: Randomized, Double Blind, Multicentric Phase III Trial Evaluating the Safety and Benefit of Adding Everolimus to Adjuvant Hormone Therapy in Women With High Risk of Relapse, ER+ and HER2- Primary Breast Cancer Who Remain Free of Disease After Receiving at Least 1 Year of Adjuvant Hormone Therapy
Brief Title: Safety Study of Adding Everolimus to Adjuvant Hormone Therapy in Women With High Risk of Relapse, ER+ and HER2- Primary Breast Cancer, Free of Disease After Receiving at Least One Year of Adjuvant Hormone Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNIRAD; 2012-003187-44 (EudraCT Number); UC-0140/1208 (Other: UNICANCER)
Record Dates: First submitted 2012-12-06; First posted 2013-03-06 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Primary Non-metastatic Breast Cancer; Who Remain Disease-free
Keywords: ER-positive HER2-negative
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Everolimus (Experimental): 1 or 2 tablets/day (i.e.5 or 10 mg/day )
  Interventions: Drug: Everolimus
- Placebo (Placebo Comparator): 1 or 2 tablets/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Everolimus — (5 or 10 mg/day, i.e. 1 or 2 tablets/day)
  Other Names: Afinitor
  Arms: Everolimus
Drug: Placebo — (5 or 10 mg/day, i.e. 1 or 2 tablets/day)
  Arms: Placebo

SUMMARY:
A significant number of patients relapse and eventually die, particularly if they were initially diagnosed with large nodes involvement and/or T3/4 diseases. When analyses focus on patients with ER+/Her2-negative breast cancer, with ≥4N+, 30% had relapsed at 5 years, emphasizing the need for new drugs in this setting (PACS01 data, UNICANCER internal data).

Strong evidence suggests that cross-talk between the phosphatidylinositol 3-kinase (PI3K)/AKT/mammalian target of rapamycin (mTOR) pathway and ER signaling is linked to hormone resistance in breast cancer patients.

In the present study, we plan to evaluate the benefit from adding everolimus to standard endocrine treatments after three years of treatment for patient ER+/HER2- at high risk of relapse due to high nodes involvement (≥4) and/or persistent node involvement after neo-adjuvant chemotherapy.

Genomic signatures have emerged during the last 10 years as a new and additive means to evaluate more precisely long term prognosis, and in some instances the amount of benefit from chemotherapy or endocrine therapy in the adjuvant setting. Therefore, the UNIRAD study can be proposed to patients with 1-3 positive lymph nodes at primary surgery and a high risk of relapse with the EndoPredict test.

This study is a unique opportunity to prove the efficacy of everolimus in adjuvant setting. The study could be practice changing in case of positive results and could allow improving outcome of breast cancer patients presenting high risk of metastatic relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Female ≥18 years of age,
2. Histologically proven invasive unilateral or bilateral breast cancer (regardless of the morphological subtype),
3. Any T, M0
4. Patient with high risk of relapse according to one of the conditions below:

   * at least 4 positive lymph nodes if the patient had primary surgery
   * or at least 1 positive lymph node if surgery was conducted after neo adjuvant chemotherapy or hormone therapy of at least 3 months duration
   * or 1-3 positive lymph nodes (pN1a, b, c) at primary surgery AND EPClin score ≥3.32867 Note: Access to primary tumor for patients with 1-3 node positive is mandatory. Patient with EPClin score <3.32867 will not be randomized, but will be followed yearly during 10 years
5. ER+ and HER2 negative : Hormone receptor positive is defined as any staining on the primary tumor, HER2 negativity is defined as IHC 0-1+, or [IHC 2+ and FISH or CISH non-amplified]
6. Primary tumor completely resected (deep margins and overlying skin involvement allowed if fully resected)
7. Patients who will begin an adjuvant hormone therapy or have received a maximum of 4 years of adjuvant hormone therapy. Hormone therapy could be either +/- LH-RH agonists, letrozole, anastrozole or exemestane.
8. No clinically or radiologically detectable metastases at time of inclusion.
9. WHO Performance status (ECOG) of 0 or 1.
10. Adequate hematological function (neutrophil count ≥2x10⁹/L; platelet count ≥ 100x10⁹/L)
11. Adequate hepatic function: AST and ALT ≤2.5 ULN, alkaline phosphatases ≤2.5 ULN, total bilirubin ≤2 ULN
12. Adequate renal function: serum creatinine ≤1.5 ULN
13. Signed written informed consent

Exclusion Criteria:

1. Any local, or regional recurrence or metastatic disease
2. Any clinical or radiological suspicion of malignant or pre-malignant disease in the contralateral breast
3. Patients with pN1mi as sole nodal involvement
4. Previous cancer (excepted basal cell carcinoma of the skin or in situ carcinoma of the cervix) in the preceding 5 years, including invasive contralateral breast cancer
5. Patient already included in another ongoing therapeutic trial involving an unlicensed drug for which follow-up is required
6. Patient who is pregnant or breast-feeding. Adequate birth control measures should be taken during the study treatment phase
7. Patient with significantly impaired lung function (e.g. Chronic Obstructive Pulmonary Disease, respiratory insufficiency, Interstitial Lung Disease)
8. Positive serology for HIV infection or hepatitis C
9. Chronic carrier of HBV (positive Antigen HbsAg positive in the blood)
10. Patient with chronic infection
11. Uncontrolled diabetes defined as glycated haemoglobin , HbA1c >7%
12. Uncontrolled hypercholesterolemia (cholesterol >300 mg/dl under adequate therapy)
13. Known hypersensitivity to the active substance, to other rapamycin derivatives or to any of the excipients
14. Patient with other concurrent severe and/or uncontrolled medical disease or infection which could compromise participation in the study (e.g. patient who regularly require systemic steroids to control co-morbid disease)
15. Patient with any psychological, familial, social or geographical condition which could potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1278 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the benefit from adding everolimus to standard endocrine treatments after two years of treatment on the disease-free survival (DFS) | 2 years

SECONDARY OUTCOMES:
Assessment of impact of everolimus on the overall survival (OS), the Event Free Survival (EFS) and Distant Metastasis Free Survival (DMFS) | 2 years
Assessment of impact of everolimus on DFS and OS in ER+,PR+ and ER+/PR- subgroups | 2 years
Impact of everolimus on the incidence of secondary cancers | 2 years
Assessment of the safety profiles for everolimus and hormone therapy combination. | 2 years
Biology: Predictive value of mTOR activation markers on DFS: IHC analysis of primary tumor for pS6K and p4EBP. | 2 years
quality of life sub-studies | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bachelot, MD, PhD, Principal Investigator — Centre Leon Berard, Lyon, France; Fabrice Andre, MD, PhD, Principal Investigator — Gustave Roussy, Villejuif, France
Locations (2):
- France (2):
  - Centre Leon Berard, Lyon
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Bidard FC, Gessain G, Bachelot T, Frechin L, Vincent-Salomon A, Drubay D, Lemonnier J, Walter T, Penault-Llorca F, Martin AL, Gaudin C, Bichat A, Sassi F, Berlemont S, Chavez-MacGregor M, Rugo HS, Badoual C, Pistilli B, Ribeiro J, Di Meglio A, Lacroix-Triki M, Vaz Luis I, Lerousseau M, Andre F. Identifying Patients With Low Relapse Rate Despite High-Risk Estrogen Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Early Breast Cancer: Development and Validation of a Clinicopathologic Assay. J Clin Oncol. 2025 Oct;43(28):3090-3101. doi: 10.1200/JCO-25-00742. Epub 2025 Aug 22. PMID 40845255
- [Derived] Giacchetti S, Laas E, Bachelot T, Lemonnier J, Andre F, Cameron D, Bliss J, Chabaud S, Hardy-Bessard AC, Lacroix-Triki M, Canon JL, Debled M, Campone M, Cottu P, Dalenc F, Ballesta A, Penault-Llorca F, Asselain B, Dumas E, Reyal F, Gougis P, Levi F, Hamy AS. Association between endocrine adjuvant therapy intake timing and disease-free survival in patients with high-risk early breast cancer: results of a sub-study of the UCBG- UNIRAD trial. EBioMedicine. 2024 Jun;104:105141. doi: 10.1016/j.ebiom.2024.105141. Epub 2024 May 7. PMID 38718683
- [Derived] Bachelot T, Cottu P, Chabaud S, Dalenc F, Allouache D, Delaloge S, Jacquin JP, Grenier J, Venat Bouvet L, Jegannathen A, Campone M, Del Piano F, Debled M, Hardy-Bessard AC, Giacchetti S, Mouret-Reynier MA, Barthelemy P, Kaluzinski L, Mailliez A, Legouffe E, Sephton M, Bliss J, Canon JL, Penault-Llorca F, Lemonnier J, Cameron D, Andre F. Everolimus Added to Adjuvant Endocrine Therapy in Patients With High-Risk Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Primary Breast Cancer. J Clin Oncol. 2022 Nov 10;40(32):3699-3708. doi: 10.1200/JCO.21.02179. Epub 2022 May 23. PMID 35605174